CLINICAL TRIAL: NCT06487962
Title: Pilot RCT: FQHC Intervention for Uptake of CGM in Low-Income Adults With T1D
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kelley Newlin Lew, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-08-011-910
Record Dates: First submitted 2024-06-13; First posted 2024-07-05 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
Keywords: Continuous Glucose Monitor; Hispanic Adult; Family; Social Ecological Model
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This study uses a mixed-methods, pragmatic pilot RCT design. Mixed-methods will be used to assess study feasibility and acceptability while quantitative methods will be used to assess RCT outcomes. As a pragmatic trial, the intervention (except peer-led support sessions) and control conditions are embedded in routine FQHC diabetes care in the participating sites.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Continuous Glucose Monitoring (CGM) Intervention Arm (Experimental): The intervention arm comprises participants receiving care from FQHC sites randomized to deliver the intervention. This arm will receive the 6-month, SEM-informed intervention to promote CGM uptake and maintenance.
  Interventions: Device: CGM Intervention
- Self-Monitoring of Blood Glucose (SMBG) Arm (Other): The SMBG control arm comprises participants receiving care from FQHC sites randomized to deliver the control condition. This arm will receive the 6-month control condition.
  Interventions: Other: SMBG Control Condition

INTERVENTIONS:
Device: CGM Intervention — The intervention has 4 components with CGM uptake and maintenance as a primary focus. (1) Participants will visit their primary care provider (PCP) at baseline and 3- and 6-months post-baseline (or more frequently as needed) for review of CGM data and insulin therapy adjustments as indicated. Intervention providers received rigorous training in T1D management and CGM via Project ECHO (Extension for Community Healthcare Outcomes). (2) After each PCP visit, the CDCES will follow-up with participants to ensure participant understanding of the education/instructions provided at the PCP visit. (3) Next, participants will receive 4-weekly sessions of culturally sensitive, intensive CGM education and training led by a CDCES with accompaniment of a supportive family member or friend. (4) Virtual group support sessions, led by a peer educator, will follow over 5 months. During this period, the peer-led sessions will take place every two weeks and then move to every three weeks.
  Arms: Continuous Glucose Monitoring (CGM) Intervention Arm
Other: SMBG Control Condition — The SMBG control condition consists of 3 components delivered over 6 months. (1) Participants will visit their PCP at baseline and 3- and 6-months post-baseline (or more frequently as needed) for review of SMBG data and insulin therapy adjustments as indicated. Control providers received rigorous training in T1D management via Project ECHO. (2) Commencing after the first PCP visit, participants will have 4-weekly telehealth visits for knowledge and skills reinforcement for SMBG. (3) CDCES support phone calls will follow over 5 months. During this period, the support phone calls will take place every two weeks and then move to every three weeks.
  Arms: Self-Monitoring of Blood Glucose (SMBG) Arm

SUMMARY:
Low-income adults with type 1 diabetes (T1D), despite their disproportionate burden of acute complications (hypoglycemia and diabetes ketoacidosis) and related emergency department visits, hospitalizations, and death, remain largely disenfranchised from continuous glucose monitoring (CGM), an efficacious technology to mitigate these inequities. To increase CGM uptake in low-income, adults with T1D receiving diabetes management in federally qualified health centers (FQHCs), this pilot randomized control trial (RCT), will assess the feasibility of our study protocol, including our multi-level intervention informed by the Socio-Ecological Model.

DETAILED DESCRIPTION:
Low-income adults with T1D experience a disproportionate burden of life-threatening, acute complications with high rates of related emergency department visits, hospitalizations, and death. Use of CGM may mitigate these inequities. Yet, low-income adults with T1D have exceptionally low levels of CGM use. This reflects social determinants of health (SODH), as framed by the multiple levels of the Socio-Ecological Model (SEM). The SEM's healthcare provider level is a main driver in Hispanic disenfranchisement from CGM. With a severe shortage of endocrinologists, primary care providers are increasingly managing T1D although many report inadequate confidence in titrating insulin and using CGM. With limited access to endocrinology, low-income, Hispanic adults with T1D thus often receive diabetes management in FQHCs with scant or no access to CGM. Hence, to foster equitable uptake of CGM in the most vulnerable adults with T1D, a 4-year, mixed-methods, feasibility study with a pilot randomized controlled trial (RCT) is underway to primarily assess the feasibility of the SEM-guided, 6-month intervention (targeting the individual, family/social networks, and healthcare provider levels). The SEM-guided intervention was refined by our Community Advisory Board. Refinements were informed by qualitative research exploring SDOH barriers to CGM uptake in low-income adults with T1D from the perspectives of four stakeholder groups.

The individual level of the intervention, guided by the Information-Motivation-Behavioral-Skills Model, fosters essential acquisition of information, motivation, and behavioral skills for CGM uptake through two principal approaches: (1) 4-week, personalized, CGM sessions with a RN/ certified diabetes care and education specialist (CDCES); and (2) subsequent virtual peer educator-led support groups, integrating CGM education, through study month six. The family/social networks level leverages social support to promote critical support in CGM uptake with a family member co-attending the 4-week sessions and participant engagement in peer-led support group sessions, respectively. The provider level of the intervention is designed to promote enhanced cultural competency in intervention delivery and provide clinical support for CGM informed by rigorous training in T1D management and CGM via Project ECHO (Extension for Community Healthcare Outcomes).

A total of 11 FQHC sites were randomized to deliver the intervention (n=6) or control (n=5) conditions with a total enrollment goal of 30 low-income adults with T1D (sites having roughly equivalent enrollment rates). The feasibility of the study protocol (e.g., recruitment and retention yields, data collection procedures, intervention implementation, and intervention acceptability, among others) will be routinely assessed. Significant intervention signals in terms of physiological (e.g., A1C and time within, above, and below range glucose range), psychosocial (e.g., quality of life and family support), and behavioral (CGM adherence) outcomes from baseline to 3- and 6-months post-baseline will be assessed. The long-term goal of this study is to inform a large, multi-site RCT, and with successful results, provide a model for CGM uptake in low-income adults with T1D for FQHCs nationally

ELIGIBILITY:
Inclusion Criteria:

* Low-income status
* Documented diagnosis of T1D
* 18 years of age or older
* Federally Qualified Health Center (FQHC) primary care provider
* English or Spanish-speaking And at intervention sites
* Willingness to wear a CGM sensor
* Adult family member or friend, who will give consent to participate in the study and co-attend the 4-week intervention sessions
* Reported difficulty in using CGM if current or past use of CGM

Exclusion Criteria:

* Pregnancy or planning to become pregnant
* Lactation
* Serious illness that may prevent study participation (e.g., severe depression)
* Less than 6 months life expectancy
* Alcohol abuse or dependence
* Uncorrected hearing or vision impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of days CGM worn | 3 months and 6 months
  The total number of days CGM worn. Data will be collected from Ambulatory Glucose Profile Reports.
Percentage of time the CGM is active | 3 months and 6 months
  The percentage of time the CGM is active. Data will be collected from Ambulatory Glucose Profile Reports.

SECONDARY OUTCOMES:
A1C | Baseline, 3 months, and 6 months
  Measure of glycemic control over the past 3 months
CGM time in range (TIR) | 3 months and 6 months
  TIR is measured by CGM. Data will be collected from Ambulatory Glucose Profile Reports.
CGM time below range (TBR) | 3 months and 6 months
  TBR is measured by CGM. Data will be collected from Ambulatory Glucose Profile Reports.
CGM time above range (TAR) | 3 months and 6 months
  TAR is measured by CGM. Data will be collected from Ambulatory Glucose Profile Reports.
Number of hypoglycemic-related emergency department (ED) visits over past 3 months | Baseline, 3 months, and 6 months
  1-item measure
Number of hypoglycemic-related hospitalizations | Baseline, 3 months, and 6 months
  1-item measure
Number of hyperglycemic-related ED visits | Baseline, 3 months, and 6 months
  1-item measure
Number of hyperglycemic-related hospitalizations | Baseline, 3 months, and 6 months
  1-item measure
Medical Outcomes Survey Short Form-36 | Baseline, 3 months, and 6 months
  Quality of Life
Multidimensional Scale of Perceived Social Support | Baseline, 3 months, and 6 months
  Social Support
Interpersonal Processes of Care Survey: Short Form | Baseline, 3 months, and 6 months
  Disparities in Interpersonal Care (communication, decision-making, and interpersonal style)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Community Health Center, Inc., Middletown, Connecticut
  - Treasure Coast Community Health, Vero Beach, Florida